CLINICAL TRIAL: NCT04925557
Title: Open-label, Single-blind, Observational, Comparative, Prospective, 36-month, Longitudinal, Controlled Study to Assess Efficacy of Siponimod (Mayzent®) on Microglia in Patients With Active Secondary Progressive Forms of Multiple Sclerosis
Brief Title: Study to Assess the Efficacy of Mayzent on Microglia in Secondary Progressive Multiple Sclerosis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director and Professor, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 00003884
Record Dates: First submitted 2021-05-24; First posted 2021-06-14 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Secondary-progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — siponimod; ocrelizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analysts had no knowledge of study drug assignment. .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrevus (Active Comparator): Patients diagnosed with secondary-progressive multiple sclerosis who have been prescribed Ocrevus by their neurologist.
  Interventions: Drug: Ocrevus
- Mayzent (Active Comparator): Patients diagnosed with secondary-progressive multiple sclerosis who have been prescribed Mayzent by their neurologist.
  Interventions: Drug: Mayzent

INTERVENTIONS:
Drug: Mayzent — PET imaging to evaluate the effects of Mayzent on the microglia of the brain.
  Arms: Mayzent
Drug: Ocrevus — PET imaging to evaluate the effects of Ocrevus on the microglia of the brain.
  Arms: Ocrevus

SUMMARY:
To assess the efficacy of Mayzent on microglia pathology in patients with active SPMS, as compared to the active control group of MS patients treated with the Ocrevus, as measured by changes in microglial activation in the lesional and non-lesional NAWM and NAGM and in the peri-plaque area of chronic lesions in the brain.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is primarily a demyelinating disease of the central nervous system (CNS), but many patients also undergo progressive atrophy, especially in the gray matter (GM). GM atrophy plays a particularly prominent role in development of cognitive and physical disability in MS. Evidence is mounting that there is a profound infiltration of activated microglia and blood-borne macrophages throughout the lesions, whereas in slowly expanding (smoldering) or chronic active expanding lesions, the microglia and macrophages are concentrated as a dense rim around the lesions. Microglia is also activated, in a more diffuse way, in the white matter (WM) and GM with concomitant axonal degeneration and meningeal inflammation. Thus, chronic activation of microglia has been linked to neurodegeneration in the progressive phase of the disease and development of brain atrophy.

No longitudinal studies in MS examined the association between development of microglia-related pathology in patients treated with siponimod (Mayzent®). This will be the first study to examine the treatment effect of Mayzent on microglia in MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with active SPMS according to the Lublin 2014 criteria. Activity is determined by MRI activity (contrast-enhancing lesions; new and unequivocally enlarging T2 lesions) and/or clinical relapses in the 24 months prior to the study baseline. If the clinical MRI is not available to determine the activity (contrast-enhancing lesions; new and unequivocally enlarging T2 lesions), then a screening MRI will be offered to the subjects to determine inclusion/exclusion criteria eligibility.
* Age between 18 and 60 years
* Have EDSS scores between 3.0 and 6.5
* Treatment naïve to both Mayzent and to Ocrevus
* Not being on S1P modulators or B-cell therapies for the last 9 months
* Subjects starting treatment as part of their clinical routine
* Be willing and able to comply with the study procedures for the duration of the trial
* Have given written informed consent and signed Health Insurance Portability and Accountability Act (HIPAA) authorization before any study-related activities are carried out
* Normal kidney functioning (creatinine clearance >59)
* No known hypersensitivity reactions to contrast agents
* None of the exclusion criteria

Exclusion Criteria:

* Have received treatment within 30 days prior to enrollment with steroids or any other concomitant immunomodulatory therapies
* Have received an investigational drug or experimental procedure within the past 30 days
* Low affinity (LAB) for the DNA single nucleotide polymorphism (SNP) of the TSPO gene on chromosome 22q13.2, using a TaqMan assay
* A CYP2C9*3/*3 genotype
* Have experienced myocardial infarction, unstable angina, stroke, TIA, decompensated heart failure requiring hospitalization, or Class III/IV heart failure in the last 6 months
* Presence of Mobitz type II second-degree, third-degree AV block, or sick sinus syndrome, unless patient has a functioning pacemaker
* Patients with active HBV confirmed by positive results for HBsAg and anti-HBV tests
* Conditions that may be associated with iron overload (e.g. hemochromatosis, thalassemia and recent blood transfusions)
* Patients with known hypersensitivity to Feraheme® or any of its components or a history of allergic reaction to any intravenous iron product
* Women who are pregnant, lactating or of childbearing age who do not consent to approved contraceptive use during the study
* Subjects who are scheduled for a routine diagnostic MRI exam in the next 4 weeks
* Other warnings and precautions to Mayzent or Ocrevus treatment according to Prescribing Information (PI) will be examined on an individual basis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo General Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with active SPMS according to the Lublin 2014 criteria. Activity is determined by MRI activity (contrast-enhancing lesions; new and unequivocally enlarging T2 lesions) and/or clinical relapses in the 24 months prior to the study baseline. Patients were recruited from 2 medical clinics.
Period: Overall Study
Arm/Group | Ocrevus | Mayzent
Started | 5 | 3
Completed | 0 (Sponsor closed the study.) | 0 (Sponsor closed the study.)
Not Completed | 5 | 3
Not completed — Study closed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Patients with relapsing remitting Multiple Sclerosis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocrevus | Mayzent | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Full Range); unit: years] | 51 [39 to 63] | 53 [49 to 55] | 52 [44 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PET Activation at 12 Months
Description: Change from baseline in PET activation of PBR06 in lesional and non-lesional NAWM and NAGM in the brain of the patients under treatment with Mayzent when 100% of patients reach 12 months;
Time Frame: 12 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in PET Activation at 6,12,24 and 36 Months Between Mayzent and Active Comparator
Description: Change from baseline in PET activation of PBR06 in lesional and non-lesional NAWM and NAGM in the brain of the patients treated with Mayzent and active control group at 6, 12, 24 and 36 months from baseline
Time Frame: 6, 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of New Ultrasmall Superparamagnetic Iron Oxide Particles
Description: The cumulative number of new ultrasmall superparamagnetic iron oxide (USPIO) particles contrast enhancing (CE) active lesions on T1-weighted images between Mayzent and active control group, as measured at 6, 12, 24 and 36 months from baseline.
Time Frame: 6, 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: MRI Measures Between Mayzent and Control-treated Groups (PBVC)
Description: Percent brain volume change (PBVC) between baseline and 12, 24, and 36 months
Time Frame: 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: MRI Measures Between Mayzent and Control-treated Groups (PCVC)
Description: Percent cortical volume change (PCVC), between baseline and 12, 24, and 36 months
Time Frame: 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: MRI Measures Between Mayzent and Control-treated Groups(PTVC)
Description: Percent thalamus volume change (PTVC) between baseline and 12, 24, and 36 months
Time Frame: 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: MRI Measures Between Mayzent and Control-treated Groups (QSM)
Description: Quantitative susceptibility mapp (QSM) change between baseline and 12, 24, and 36 months
Time Frame: 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Cumulative Number of New Gadolinium CE Lesions
Description: The cumulative number of new gadolinium CE lesions on T1-weighted images at months 6, 12, 24 and 36 months
Time Frame: 6, 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Cumulative Number of New or Newly Enlarging T2 Lesions
Description: The cumulative number of new or newly enlarging hyperintense T2 lesions measured at months 6, 12, 24 and 36 months
Time Frame: 6, 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Absolute Change in Hyperintense T2 Lesions Volume
Description: The absolute change in hyperintense T2-lesion volume (LV) measured at months 6, 12, 24 and 36 months
Time Frame: 6, 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Absolute Change in Hypo-intense T1 Lesions Volume
Description: The absolute change in hypo-intense T1-lesion volume (LV) measured at months 6, 12, 24 and 36 months
Time Frame: 6, 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Absolute Change in Serum Neurofilament and Glial Protein
Description: The absolute change in serum neurofilament light chain (sNfL) and glial fibrillary acidic protein (GFAP) at 6, 12, 24 and 36 months
Time Frame: 6, 12, 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Association Between Imaging and Clinical and Cognitive Outcomes
Description: The association between imaging and clinical and cognitive outcomes, incl. the composite EDSS+SDMT, over 24 and 36 months of the study
Time Frame: 24 and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Number of Participants With Treatment Related Adverse Events
Description: Safety of Mayzent and active control group over 12, 24, and 36 months of the study
Time Frame: 12, 24, and 36 months
Population: Study was terminated. No subject had any further data collected after the initial visit.
Arm/Group | Ocrevus | Mayzent
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 5 months.
Description: Case form provided by the study sponsor.
Arm/Group | Ocrevus | Mayzent
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrevus (N=5) | Mayzent (N=3)
Allergic Reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) — Fever, chills, headache, numbness in face.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04925557/Prot_SAP_ICF_000.pdf